CLINICAL TRIAL: NCT03150927
Title: A Clinical Study to Determine the Effects of a Novel Probiotic Microbial Composite™ on Improving Digestive Health and Key Growth Parameters in Undernourished Young Children
Brief Title: Clinical Study of Novel Probiotic Microbial Composite™ to Treat Undernourished Young Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biowish Technologies, Inc. (Other)
Collaborators: University of Wollongong (Other); Mysore Medical College and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BWT-20150720-001
Record Dates: First submitted 2017-04-05; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Quality of Life; Malnutrition; Growth Arrest
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: The Randomized Clinical Trial (RCT) will typically involve 250 subjects randomized into two arms based on age and sex.
  Following a positive outcome in the RCT (following 6 months), we envisage converting the study to an observational based study (case-study) based on ethical principles where the placebo arm of the study would be administered the test product. Each subject will be assessed for a total of two years.
Who Masked: Participant, Care Provider
Masking Description: Product will be given to subjects in a capsule form. Participant and participants legal guardians, and care providers will not know if the capsule is a placebo or the Probiotic Microbial Composite™
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Microbial Composite (Experimental): Probiotic Microbial Composite is a safe, 100% natural material containing all Generally Recognized as Safe (GRAS) Probiotics, combined with FDA approved food grade excipient materials. The probiotics contained within are also all 100% natural and non-Genetically Modified Organisms (non-GMO).
  Interventions: Dietary Supplement: Probiotic Microbial Composite
- Placebo (Placebo Comparator): Placebo is a mixture of inactive ingredients found in Probiotic Microbial Composite. These ingredients are FDA approved food grade materials, 100% natural and palatable.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Microbial Composite — 125mg (or 250 mg) of BiOWiSH Probiotic Microbial Composite™ is to be dosed once daily. Product will be supplied in capsule form to be administered orally. Each subject will be given a 15-day supply (30 capsules) to take with them after their initial visit. Capsules will be administered every 15 days by primary investigators at follow up visits.
  Arms: Probiotic Microbial Composite
Dietary Supplement: Placebo — 125mg (or 250 mg) of Placebo is to be dosed once daily. Product will be supplied in capsule form to be administered orally. Each subject will be given a 15-day supply (30 capsules) to take with them after their initial visit. Capsules will be administered every 15 days by primary investigators at follow up visits.
  Arms: Placebo

SUMMARY:
This study is to determine if a novel bio-fermented Microbiotic Composite™ can improve the digestive health and subsequent growth and quality of life parameters in a selected group of children in a district in India.

DETAILED DESCRIPTION:
The Probiotic Microbial Composite™ is a multifaceted technology that encompasses three key areas, namely, prebiotics, probiotics and post-biotics. The first component, prebiotics, involve non-digestible food ingredients, typically oligosaccharides which act by beneficially affecting the host by stimulating growth, activity, or in fact both of specific intestinal bacteria.

The probiotic component refers to the augmentation or addition of bacteria to enhance and support the various beneficial bacteria that are inherent to the gastrointestinal tract. The bio-fermented Microbiotic Composite™ is a consortium of bacteria which can play a significant physiological role as a probiotic. This theory, termed the microbial consortium theory suggests that rather than a cumulative effect by the bacteria, there is in fact combinatorial affect by the use of several species.

The final component post-biotics, in general, mimic the beneficial health promoting effects of probiotics whilst avoiding the risk of taking live micro-organisms within the gastrointestinal tract, especially in populations such as infants and the elderly in whom the intestinal barriers, as well as, innate immune defenses can be impaired. The term typically encompasses a vast plethora of byproducts, know as metabolites, produced and secreted by the bacteria in response to their environment.

ELIGIBILITY:
The Randomized Clinical Trial (RCT) will typically involve 250 subjects randomized into two arms based on age and sex.

Following a positive outcome in the RCT (following 6 months), we envisage converting the study to an observational based study (case-study) based on ethical principles where the placebo arm of the study would be administered the test product. Each subject will be assessed for a total of two years.

Inclusion criteria:

* Inpatient setting: Children with age of 3 years to 12 years with acute diarrhea
* Outpatient setting: healthy children aged 3 years to 12 years

Exclusion criteria:

* Subjects taking any kind of prescription medication.
* Subjects taking any dietary supplements (2-week washout is permitted).
* Subjects taking any antibiotics (must have discontinued antibiotic use 12-weeks prior to beginning study). An allowance will be made to existing subjects already taking part in the study. This confounder will however have to be noted by the primary investigators.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

  * Including subjects who are bed or wheelchair-bound
  * Including subjects who have any physical disability which could interfere with their ability to perform the functional performance measures included in this protocol.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Acute diarrhea in children ages 3 years to 12 years | 24 weeks
  Subjects will be assessed as to severity of diarrhea using a standardized measure of diarrheal severity in pediatrics

SECONDARY OUTCOMES:
Serial assessment of healthy children aged 3 years to 12 years | 2 years
  Subjects will be followed by serial assessment of mid-arm circumference measured in centimeters.
Serial assessment of healthy children aged 3 years to 12 years | 2 years
  Subjects will be followed by serial assessment of head circumference measured in centimeters.
Height of healthy children aged 3 years to 12 years | 2 years
  Subjects will be followed by serial assessment of height in centimeters
Weight of healthy children aged 3 years to 12 years | 2 years
  Subjects will be followed by serial assessment of weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Mudassir A Khan, Ph.D., Principal Investigator — Department of Community Medicine/Public Health Mysore Medical College & Research Institute; Amit Kapur, MBBS, Principal Investigator — Prince of Wales Hospital; Richard S Carpenter, PhD, Principal Investigator — Biowish Technologies, Inc.
Locations (1):
- Mysore Medical College and Research Institute, Mysore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allen SJ, Okoko B, Martinez E, Gregorio G, Dans LF. Probiotics for treating infectious diarrhoea. Cochrane Database Syst Rev. 2004;(2):CD003048. doi: 10.1002/14651858.CD003048.pub2. PMID 15106189
- [Background] Asuzu MC. A comparative study of the commonly used nutritional assessment tools for primary health care. East Afr Med J. 1991 Nov;68(11):913-22. PMID 1800086
- [Background] Bhutta ZA, Das JK. Interventions to address maternal and childhood undernutrition: current evidence. Nestle Nutr Inst Workshop Ser. 2014;78:59-69. doi: 10.1159/000354941. Epub 2014 Jan 27. PMID 24504207
- [Background] Canani RB, Cirillo P, Terrin G, Cesarano L, Spagnuolo MI, De Vincenzo A, Albano F, Passariello A, De Marco G, Manguso F, Guarino A. Probiotics for treatment of acute diarrhoea in children: randomised clinical trial of five different preparations. BMJ. 2007 Aug 18;335(7615):340. doi: 10.1136/bmj.39272.581736.55. Epub 2007 Aug 9. PMID 17690340
- [Background] D'Souza AL, Rajkumar C, Cooke J, Bulpitt CJ. Probiotics in prevention of antibiotic associated diarrhoea: meta-analysis. BMJ. 2002 Jun 8;324(7350):1361. doi: 10.1136/bmj.324.7350.1361. PMID 12052801
- [Background] Depeint F, Tzortzis G, Vulevic J, I'anson K, Gibson GR. Prebiotic evaluation of a novel galactooligosaccharide mixture produced by the enzymatic activity of Bifidobacterium bifidum NCIMB 41171, in healthy humans: a randomized, double-blind, crossover, placebo-controlled intervention study. Am J Clin Nutr. 2008 Mar;87(3):785-91. doi: 10.1093/ajcn/87.3.785. PMID 18326619
- [Background] Fang SB, Lee HC, Hu JJ, Hou SY, Liu HL, Fang HW. Dose-dependent effect of Lactobacillus rhamnosus on quantitative reduction of faecal rotavirus shedding in children. J Trop Pediatr. 2009 Oct;55(5):297-301. doi: 10.1093/tropej/fmp001. Epub 2009 Feb 8. PMID 19203988
- [Background] Grosse SD, Roy K. Long-term economic effect of early childhood nutrition. Lancet. 2008 Feb 2;371(9610):365-6. doi: 10.1016/S0140-6736(08)60180-4. No abstract available. PMID 18242398
- [Background] Guarino A, Canani RB, Spagnuolo MI, Albano F, Di Benedetto L. Oral bacterial therapy reduces the duration of symptoms and of viral excretion in children with mild diarrhea. J Pediatr Gastroenterol Nutr. 1997 Nov;25(5):516-9. doi: 10.1097/00005176-199711000-00005. PMID 9360205
- [Background] Gueimonde M, Sakata S, Kalliomaki M, Isolauri E, Benno Y, Salminen S. Effect of maternal consumption of lactobacillus GG on transfer and establishment of fecal bifidobacterial microbiota in neonates. J Pediatr Gastroenterol Nutr. 2006 Feb;42(2):166-70. doi: 10.1097/01.mpg.0000189346.25172.fd. PMID 16456409
- [Background] Hoddinott J, Maluccio JA, Behrman JR, Flores R, Martorell R. Effect of a nutrition intervention during early childhood on economic productivity in Guatemalan adults. Lancet. 2008 Feb 2;371(9610):411-6. doi: 10.1016/S0140-6736(08)60205-6. PMID 18242415
- [Background] Hooper LV, Midtvedt T, Gordon JI. How host-microbial interactions shape the nutrient environment of the mammalian intestine. Annu Rev Nutr. 2002;22:283-307. doi: 10.1146/annurev.nutr.22.011602.092259. Epub 2002 Apr 4. PMID 12055347
- [Background] Johnston BC, Supina AL, Ospina M, Vohra S. Probiotics for the prevention of pediatric antibiotic-associated diarrhea. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD004827. doi: 10.1002/14651858.CD004827.pub2. PMID 17443557
- [Background] Kalliomaki M, Salminen S, Poussa T, Isolauri E. Probiotics during the first 7 years of life: a cumulative risk reduction of eczema in a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2007 Apr;119(4):1019-21. doi: 10.1016/j.jaci.2006.12.608. Epub 2007 Feb 7. No abstract available. PMID 17289135
- [Background] Kosek M, Bern C, Guerrant RL. The global burden of diarrhoeal disease, as estimated from studies published between 1992 and 2000. Bull World Health Organ. 2003;81(3):197-204. Epub 2003 May 16. PMID 12764516
- [Background] Laparra JM, Sanz Y. Comparison of in vitro models to study bacterial adhesion to the intestinal epithelium. Lett Appl Microbiol. 2009 Dec;49(6):695-701. doi: 10.1111/j.1472-765X.2009.02729.x. Epub 2009 Aug 25. PMID 19843211
- [Background] Laparra JM, Sanz Y. Interactions of gut microbiota with functional food components and nutraceuticals. Pharmacol Res. 2010 Mar;61(3):219-25. doi: 10.1016/j.phrs.2009.11.001. Epub 2009 Nov 13. PMID 19914380
- [Background] Lefkovitz AL, Zarowitz BJ. It's a microscopic world after all: prebiotics, probiotics, and synbiotics. Geriatr Nurs. 2013 Jul-Aug;34(4):323-5. doi: 10.1016/j.gerinurse.2013.06.007. No abstract available. PMID 23916327
- [Background] Marteau P, Shanahan F. Basic aspects and pharmacology of probiotics: an overview of pharmacokinetics, mechanisms of action and side-effects. Best Pract Res Clin Gastroenterol. 2003 Oct;17(5):725-40. doi: 10.1016/s1521-6918(03)00055-6. PMID 14507584
- [Background] Mountzouris KC, McCartney AL, Gibson GR. Intestinal microflora of human infants and current trends for its nutritional modulation. Br J Nutr. 2002 May;87(5):405-20. doi: 10.1079/BJNBJN2002563. PMID 12010580
- [Background] Owen GM. The new National Center for Health Statistics growth charts. South Med J. 1978 Mar;71(3):296-7. doi: 10.1097/00007611-197803000-00027. No abstract available. PMID 628854
- [Background] Patel RM, Denning PW. Therapeutic use of prebiotics, probiotics, and postbiotics to prevent necrotizing enterocolitis: what is the current evidence? Clin Perinatol. 2013 Mar;40(1):11-25. doi: 10.1016/j.clp.2012.12.002. Epub 2013 Jan 17. PMID 23415261
- [Background] Pedone CA, Arnaud CC, Postaire ER, Bouley CF, Reinert P. Multicentric study of the effect of milk fermented by Lactobacillus casei on the incidence of diarrhoea. Int J Clin Pract. 2000 Nov;54(9):568-71. PMID 11220983
- [Background] Pedone CA, Bernabeu AO, Postaire ER, Bouley CF, Reinert P. The effect of supplementation with milk fermented by Lactobacillus casei (strain DN-114 001) on acute diarrhoea in children attending day care centres. Int J Clin Pract. 1999 Apr-May;53(3):179-84. PMID 10665128
- [Background] Ruemmele FM, Bier D, Marteau P, Rechkemmer G, Bourdet-Sicard R, Walker WA, Goulet O. Clinical evidence for immunomodulatory effects of probiotic bacteria. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):126-41. doi: 10.1097/MPG.0b013e31817d80ca. PMID 19179874
- [Background] Saavedra JM, Bauman NA, Oung I, Perman JA, Yolken RH. Feeding of Bifidobacterium bifidum and Streptococcus thermophilus to infants in hospital for prevention of diarrhoea and shedding of rotavirus. Lancet. 1994 Oct 15;344(8929):1046-9. doi: 10.1016/s0140-6736(94)91708-6. PMID 7934445
- [Background] Sanz Y, De Palma G. Gut microbiota and probiotics in modulation of epithelium and gut-associated lymphoid tissue function. Int Rev Immunol. 2009;28(6):397-413. doi: 10.3109/08830180903215613. PMID 19954356
- [Background] Schoeman SE, Hendricks MK, Hattingh SP, Benade AJ, Laubscher JA, Dhansay MA. The targeting of nutritionally at-risk children attending a primary health care facility in the Western Cape Province of South Africa. Public Health Nutr. 2006 Dec;9(8):1007-12. doi: 10.1017/s1368980006009864. PMID 17125564
- [Background] Schwiertz A, Gruhl B, Lobnitz M, Michel P, Radke M, Blaut M. Development of the intestinal bacterial composition in hospitalized preterm infants in comparison with breast-fed, full-term infants. Pediatr Res. 2003 Sep;54(3):393-9. doi: 10.1203/01.PDR.0000078274.74607.7A. Epub 2003 Jun 4. PMID 12788986
- [Background] Shanahan F. Probiotics: a perspective on problems and pitfalls. Scand J Gastroenterol Suppl. 2003;(237):34-6. doi: 10.1080/00855910310001476. PMID 12797679
- [Background] Szajewska H, Mrukowicz J. Meta-analysis: non-pathogenic yeast Saccharomyces boulardii in the prevention of antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2005 Sep 1;22(5):365-72. doi: 10.1111/j.1365-2036.2005.02624.x. PMID 16128673
- [Background] Szajewska H, Ruszczynski M, Radzikowski A. Probiotics in the prevention of antibiotic-associated diarrhea in children: a meta-analysis of randomized controlled trials. J Pediatr. 2006 Sep;149(3):367-372. doi: 10.1016/j.jpeds.2006.04.053. PMID 16939749
- [Background] Szajewska H, Skorka A, Dylag M. Meta-analysis: Saccharomyces boulardii for treating acute diarrhoea in children. Aliment Pharmacol Ther. 2007 Feb 1;25(3):257-64. doi: 10.1111/j.1365-2036.2006.03202.x. PMID 17269987
- [Background] Tlaskalova-Hogenova H, Stepankova R, Hudcovic T, Tuckova L, Cukrowska B, Lodinova-Zadnikova R, Kozakova H, Rossmann P, Bartova J, Sokol D, Funda DP, Borovska D, Rehakova Z, Sinkora J, Hofman J, Drastich P, Kokesova A. Commensal bacteria (normal microflora), mucosal immunity and chronic inflammatory and autoimmune diseases. Immunol Lett. 2004 May 15;93(2-3):97-108. doi: 10.1016/j.imlet.2004.02.005. PMID 15158604
- [Background] Tsilingiri K, Rescigno M. Postbiotics: what else? Benef Microbes. 2013 Mar 1;4(1):101-7. doi: 10.3920/BM2012.0046. PMID 23271068
- [Background] Weizman Z, Asli G, Alsheikh A. Effect of a probiotic infant formula on infections in child care centers: comparison of two probiotic agents. Pediatrics. 2005 Jan;115(1):5-9. doi: 10.1542/peds.2004-1815. PMID 15629974
- [Background] Wingreen NS, Levin SA. Cooperation among microorganisms. PLoS Biol. 2006 Sep;4(9):e299. doi: 10.1371/journal.pbio.0040299. PMID 16968138
- [Background] Zoetendal EG, Rajilic-Stojanovic M, de Vos WM. High-throughput diversity and functionality analysis of the gastrointestinal tract microbiota. Gut. 2008 Nov;57(11):1605-15. doi: 10.1136/gut.2007.133603. PMID 18941009
- [Background] Borody TJ, Peattie D, Kapur A. Could fecal microbiota transplantation cure all Clostridium difficile infections? Future Microbiol. 2014;9(1):1-3. doi: 10.2217/fmb.13.146. No abstract available. PMID 24328373
- [Background] Cremonini F, Di Caro S, Nista EC, Bartolozzi F, Capelli G, Gasbarrini G, Gasbarrini A. Meta-analysis: the effect of probiotic administration on antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2002 Aug;16(8):1461-7. doi: 10.1046/j.1365-2036.2002.01318.x. PMID 12182746
- [Background] Cunliffe NA, Kilgore PE, Bresee JS, Steele AD, Luo N, Hart CA, Glass RI. Epidemiology of rotavirus diarrhoea in Africa: a review to assess the need for rotavirus immunization. Bull World Health Organ. 1998;76(5):525-37. PMID 9868844
- [Background] Dabek M, McCrae SI, Stevens VJ, Duncan SH, Louis P. Distribution of beta-glucosidase and beta-glucuronidase activity and of beta-glucuronidase gene gus in human colonic bacteria. FEMS Microbiol Ecol. 2008 Dec;66(3):487-95. doi: 10.1111/j.1574-6941.2008.00520.x. Epub 2008 Jun 4. PMID 18537837
- [Background] Dubey AP, Rajeshwari K, Chakravarty A, Famularo G. Use of VSL[sharp]3 in the treatment of rotavirus diarrhea in children: preliminary results. J Clin Gastroenterol. 2008 Sep;42 Suppl 3 Pt 1:S126-9. doi: 10.1097/MCG.0b013e31816fc2f6. PMID 18806703
- [Background] Gronlund MM, Lehtonen OP, Eerola E, Kero P. Fecal microflora in healthy infants born by different methods of delivery: permanent changes in intestinal flora after cesarean delivery. J Pediatr Gastroenterol Nutr. 1999 Jan;28(1):19-25. doi: 10.1097/00005176-199901000-00007. PMID 9890463
- [Background] Hapfelmeier S, Lawson MA, Slack E, Kirundi JK, Stoel M, Heikenwalder M, Cahenzli J, Velykoredko Y, Balmer ML, Endt K, Geuking MB, Curtiss R 3rd, McCoy KD, Macpherson AJ. Reversible microbial colonization of germ-free mice reveals the dynamics of IgA immune responses. Science. 2010 Jun 25;328(5986):1705-9. doi: 10.1126/science.1188454. PMID 20576892
- [Background] International Conference on Primary Health Care. Declaration of Alma-Ata. WHO Chron. 1978 Nov;32(11):428-30. No abstract available. PMID 11643481
- [Background] Johnson CL, Versalovic J. The human microbiome and its potential importance to pediatrics. Pediatrics. 2012 May;129(5):950-60. doi: 10.1542/peds.2011-2736. Epub 2012 Apr 2. PMID 22473366
- [Background] Kawamoto S, Tran TH, Maruya M, Suzuki K, Doi Y, Tsutsui Y, Kato LM, Fagarasan S. The inhibitory receptor PD-1 regulates IgA selection and bacterial composition in the gut. Science. 2012 Apr 27;336(6080):485-9. doi: 10.1126/science.1217718. PMID 22539724
- [Background] Rautava S, Arvilommi H, Isolauri E. Specific probiotics in enhancing maturation of IgA responses in formula-fed infants. Pediatr Res. 2006 Aug;60(2):221-4. doi: 10.1203/01.pdr.0000228317.72933.db. PMID 16864708
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867